CLINICAL TRIAL: NCT06919120
Title: The Study on the Effect of Different Administration Methods of Simethicone in Reducing Bubbles During Bowel Preparation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: KY-2024-227
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-12

CONDITIONS: Colonoscopy
Keywords: Dimethicone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): The patients in this group mixed one bottle of simethicone into the final packet of compound polyethylene glycol electrolyte powder, dissolved it in 1000 ml of water, and consumed it within one hour.
  Interventions: Drug: Simethicone is mixed into the final packet of compound polyethylene glycol electrolyte powder
- B (Experimental): The patients in this group took one bottle of simethicone orally after finishing the last sip of compound polyethylene glycol electrolyte solution.
  Interventions: Drug: Take simethicone separately

INTERVENTIONS:
Drug: Simethicone is mixed into the final packet of compound polyethylene glycol electrolyte powder — The patients added one bottle of simethicone when taking the final packet of compound polyethylene glycol electrolyte powder.
  Arms: A
Drug: Take simethicone separately — Take one bottle of simethicone orally after finishing the last sip of compound polyethylene glycol electrolyte solution.
  Arms: B

SUMMARY:
To find the simplest and most effective method of intestinal preparation for dimethicone administration.

DETAILED DESCRIPTION:
A randomized controlled trial of dimethicone mixed with compound polyethylene glycol electrolyte powder (group A) versus dimethicone alone was conducted in patients undergoing colonoscopy (group B) the two different administration methods were used to compare the defoaming effect of dimethicone and the detection rate of polyps ≤0.5cm. To find the best way to administer dimethicone during bowel preparation for colonoscopy.

In group A (n = 686), a bottle of dimethicone was mixed with the last package of compound polyethylene glycol electrolyte powder, dissolved in 1000ml water, and finished within 1 hour during bowel preparation.

Group B (n = 686) received a bottle of dimethicone after taking the last sip of compound polyethylene glycol electrolyte powder.

Investigators asked each patient and physician about the interval between the administration of dimethicone and the initiation of colonoscopy, the time to colonoscopy withdrawal, the bowel cleanliness score, the intestinal bubble score, and whether polyps ≤0.5cm in diameter were detected.

SPSS25.0 was used to analyze the data with two independent samples t test. The gender, age, the interval between the end of antifoams and the start of the examination, the time of withdrawal from colonoscopy during the examination, the intestinal cleanliness score, the intestinal bubble score, and the detection of polyps with diameter ≤0.5cm were analyzed between group A (dimethicone mixed with compound polyethylene glycol electrolyte powder) and group B (dimethicone alone).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine colonoscopy at our hospital are aged between 18 to 80 years, including those who meet the Indications for colonoscopy without any absolute contraindications.

Exclusion Criteria:

* （１） suffering from pancoliنى, intestinal obstruction, toxic megacolon, severe acute gastrointestinal infection, etc.; （２） individuals with severe dysfunction of the heart, lungs, liver, kidneys, etc.; （３） individuals with a history of allergic reaction to the above gastrointestinal agents; （４） individuals who cannot consent to treatment for epilepsy, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | During the colonoscopy procedure
  Bowel cleanliness was assessed using the Boston Bowel Preparation Scale (BBPS) in both groups, and the efficacy of bowel cleansing was compared between the two medication regimens to identify potential differences
Intestinal Bubble Score | During the colonoscopy procedure
  Bowel foam levels were assessed using the Intestinal Bubble Score (IBS) in both groups, and the efficacy of foam clearance was compared between the two medication regimens to identify potential differences

SECONDARY OUTCOMES:
Detection rate of polyps | During the colonoscopy procedure
  The detection rate of polyps ≤0.5 cm was compared between the two groups

OTHER OUTCOMES:
Time taken for colonoscope withdrawal | During the colonoscopy procedure
  Record the endoscopy retraction time for two groups and compare whether there is a difference in the retraction time of endoscopy under the two different medication regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Affiliated Hospital of Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided